CLINICAL TRIAL: NCT03746691
Title: Effect of Citalopram on Fasting and Postprandial Lower Esophageal Sphincter Function in Healthy Subjects: a Double-blind, Placebo-controlled, Randomized, Cross-over Study
Brief Title: Effect of Citalopram on Reflux Episodes in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S59148
Record Dates: First submitted 2017-03-21; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citalopram, 20 mg, IV (Experimental): After placement of a high resolution impedance manometry catheter (transnasally), citalopram will be administered IV over 30 minutes (20 mg in 100ml saline). Thereafter, the investigators will wait for 20 minutes, after which the volunteers will receive 10 wet swallows (5ml saline), to investigate esophageal peristalsis. Thereafter, a standard meal (1000kcal) will be given to the volunteers and recordings will continue for another 2 hours.
  Interventions: Drug: Citalopram HCl
- Placebo, IV (Placebo Comparator): After placement of a high resolution impedance manometry catheter (transnasally), placebo (saline 100ml) will be administered IV over 30 minutes. Thereafter, the investigators will wait for 20 minutes, after which the volunteers will receive 10 wet swallows (5ml saline), to investigate esophageal peristalsis. Thereafter, a standard meal (1000kcal) will be given to the volunteers and recordings will continue for another 2 hours.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Citalopram HCl — Citalopram HCl IV 20 mg in 100 ml saline will be infused IV over the course of 30 minutes. Volunteers will receive a standard meal, and recordings using high resolution impedance manometry, will be continued for 2 hours.
  Arms: Citalopram, 20 mg, IV
Drug: Placebos — Placebo (100 ml saline IV) will be infused IV over the course of 30 minutes. Volunteers will receive a standard meal, and recordings using high resolution impedance manometry, will be continued for 2 hours.
  Arms: Placebo, IV

SUMMARY:
Citalopram is sometimes used in the treatment for gastro-esophageal reflux disease, however, there are no empirical data to support this. The investigators would like to know if citalopram has an effect on the lower esophageal sphincter pressure, transient lower esophageal sphincter relaxations and reflux episodes. The investigators will investigate this by performing high resolution impedance manometry in healthy volunteers before and after a solid meal. This will be compared to placebo, in a cross-over, randomized, double-blind condition.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years

Exclusion Criteria:

* history of upper GI symptoms
* history of upper GI surgery
* psychological disorders
* any drug history
* use of medication altering GI motility
* nursing and pregnant woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in LES pressure | LES pressure will be measured for 4 times (a 5 sec time window) per hour. The average of the first hour will be taken as the LES pressure for the first hour postprandially.
  The investigators will measure lower esophageal sphincter pressure after a meal between placebo and citalopram, using a high resolution impedance manometry system. LES pressures will be measured in the first hour postprandial and will be compared (preprandial vs postprandial hour 1).
Change in the number of reflux episodes | The number of reflux episodes will be counted in a 3 hour time period, to have 1 number of reflux episodes.
  The investigators will measure the number of reflux episodes after a meal between placebo and citalopram, using a high resolution impedance manometry system.
Change in the number of TLESRs | The total number of TLESRs will be counted in a 3 hour time period, to have 1 number of TLESRs.
  The investigators will measure the number of transient lower esophageal sphincter relaxations after a meal between placebo and citalopram, using a high resolution impedance manometry system.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided